CLINICAL TRIAL: NCT00012779
Title: Effectiveness of a Health Education Program in a Primary Care Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 95-118
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-06

CONDITIONS: Frail Elderly
Keywords: Health Care Education; Health Care Cost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: Health Education Program

SUMMARY:
This study was designed to assess the effectiveness of a Health Education Program (HEP) for improving the well-being and reducing the health care use and cost of care of frail older outpatient veterans, and for improving the well-being of their spouse caregivers. HEP is a multi-component group program delivered in 8 weekly, 2-hour sessions, and 10 monthly 2-hour follow-up sessions, it includes emotion-focused and problem focused coping strategies, education and support.

DETAILED DESCRIPTION:
Background:

This study was designed to assess the effectiveness of a Health Education Program (HEP) for improving the well-being and reducing the health care use and cost of care of frail older outpatient veterans, and for improving the well-being of their spouse caregivers. HEP is a multi-component group program delivered in 8 weekly, 2-hour sessions, and 10 monthly 2-hour follow-up sessions, it includes emotion-focused and problem focused coping strategies, education and support.

Objectives:

The objectives of this study are to evaluate: 1) effects of HEP on the perceived health status, emotional well-being, and social support of frail veterans; 2) effects of HEP on the perceived health, emotional well-being, social support, burden levels, self-appraisal of change, pressing problems associated with caregiving, knowledge and use of community resources by caregiver; and 3) effects of HEP on the health care use and costs of care recipients.

Methods:

HEP was evaluated using a randomized control group design. The design has two levels of intervention, HEP vs. Usual Care (UC), 3 VA medical centers (VAMCs), and 4 times of measurement (at baseline, after the 8th HEP meeting, and at 1 and 2 years after baseline). Data reported here are for 8 week and 1-year psychosocial outcomes and 18 months for VA cost. Caregivers and veterans (n = 466) were randomized in 3 VAMCs, 114 to UC and 119 to HEP. The typical caregiver was 68 years old, married, white, female, with some college education and living with the veteran. The typical veteran care recipient was 74 years old, white, male with some college education, and suffered from one or more chronic health problems. Fifteen HEP groups were conducted. Caregivers and recipients were assessed on: 1) health and functional status; 2) emotional well-being; and 3) social support. In addition, caregivers were assessed for change in coping skills, change in burden level, pressing problems, and knowledge and use of community resources. Data was analyzed using random effects regression models.

Status:

Data on two-year outcomes for health and functional status, emotional well-being, and social support of caregivers and veterans, problems associated with caregiving and Medicare plus VA costs are being collected and analyzed for an amended final report.

ELIGIBILITY:
Inclusion Criteria:

Caregiver inclusion criteria: 2) married to, and living with, the care recipient; 2) age 55 and older; 3) being the primary care provider for the care recipient and reporting at least a moderate level of burden on the Caregiver Strain Index; 4) report spouse has poor health care; and 5) receiver age 55 and suffering from chronic health condition.

Exclusion Criteria:

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B. Engelhardt, PhD, Principal Investigator — Albany VA Medical Center Samuel S. Stratton, Albany, NY
Locations (3):
- United States (3):
  - VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts
  - Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York